CLINICAL TRIAL: NCT05503381
Title: A Randomized, Controlled, Multicenter, Noninferiority Study of Perioperative and Oncological Safety of Transanal Laparoscopic Radical Resection of Low Rectal Cancer (NOSES I) Compared With Conventional Laparoscopic Assisted Surgery for Low Rectal Cancer
Brief Title: A Randomized, Controlled, Multicenter, Noninferiority Clinical Study of Perioperative and Oncological Safety in Patients With Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhenglou, Associate chief physician and associate professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-NOSES
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Department of Anorectal Surgery, Changhai Hospital Affiliated to Naval Medical University
Keywords: Colorectal cancer；Natural Orifice Specimen Extraction Surgery；Disease-free survival

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, multicenter, noninferiority clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Orifice Specimen Extraction Surgery Group (Experimental): The patient underwent laparoscopic lower rectal cancer surgery with transanal specimen collection
  Interventions: Procedure: Laparoscopic radical resection of low rectal cancer with transanal specimens
- Traditional laparoscopic surgery (No Intervention): The patient underwent conventional laparoscopic lower rectal cancer surgery

INTERVENTIONS:
Procedure: Laparoscopic radical resection of low rectal cancer with transanal specimens — According to the standard laparoscopic anterior rectum resection, the rectum was separated 2-3cm below the tumor, the rectum was severed 1-2cm from the lower edge of the tumor, the rectal stump was connected with the tumor through the anus, and the sigmoid colon was severed 10cm from the upper edge of the tumor. The stapler head was placed in the sigmoid colon stump, and then the sigmoid colon stump was closed with a linear cutting closure device. Then, the sigmoid colon stump is returned to the abdominal cavity through the anus, the distal rectal stump is closed with a suture purse or a linear cutting closure device, and the stapler body is inserted through the anus, and then the anastomosis is completed.
  Arms: Natural Orifice Specimen Extraction Surgery Group

SUMMARY:
Laparoscopic natural orifice specimen extraction surgery (NOSES) for low rectal cancer has a good minimally invasive effect. However, the NOSES prognosis studies are all small sample retrospective studies. This study conducted a multicenter prospective randomized controlled trial of NOSES surgery for low rectal cancer to compare the difference in surgical outcomes between conventional laparoscopic surgery and NOSES surgery for low rectal cancer. A total of 500 patients were planned to be enrolled, including 250 in the control group and 250 in the experimental group. The primary end point was 2-year disease-free survival (DFS), and the secondary end points were surgical safety, postoperative pathology, postoperative defecation, urination, and sexual function. Through a large sample size study, this study aims to clarify the advantages of NOSE surgery for low rectal cancer, promote the promotion of low rectal cancer NOSES surgery in the country, standardize the way of low rectal cancer NOSES surgery, improve the surgical treatment of patients with low rectal cancer, improve the quality of life of patients, reduce the burden of patients, and increase the satisfaction. And improve the international influence of the project team in the field of minimally invasive surgical treatment of colorectal cancer.

DETAILED DESCRIPTION:
Research Objectives:

1. To compare the difference in the oncological effect between laparoscopic radical resection of low rectal cancer with anal specimens (NOSES I type) and laparoscopic assisted surgery for low rectal cancer;
2. To compare the safety of laparoscopic radical resection of low rectal cancer with anal specimens (NOSES I type) and laparoscopic assisted surgery for low rectal cancer within 30 days of perioperative period;
3. To explore the difference in the prophylactic stoma implementation and the positive rate of tumor cells in pelvic flushing fluid between laparoscopic radical resection of low rectal cancer with anal specimens (NOSES I) and laparoscopic assisted resection of lower rectal cancer.

Primary end Point: 2-year Disease-free survival (DFS) Secondary end points :(1) incidence of SSI; (2) Incidence of serious postoperative complications (anastomotic leakage, postoperative bleeding, etc.); (3) R0 removal rate; (4) Postoperative recovery (pain, exhaust and defecation time, eating time, postoperative hospital stay, etc.); (5) Postoperative pathological conditions (distance between upper and lower margins, number of lymph nodes, circumferential margins, etc.); (6) 2-year RFS and OS.

Exploratory end points :(1) prophylactic colostomy rate; (2) Positive rate of tumor cells in pelvic flushing fluid.

Inclusion criteria:

1. Patients aged 18-75 years;
2. Adenocarcinoma confirmed by pathology;
3. colonoscopy or imaging examination confirmed that the distance between the lower edge of the tumor and the anal edge was less than 5cm;
4. Preoperative imaging diagnosis was CT1-3NXM0;
5. Preoperative colonoscopy or imaging diagnosis confirmed that the maximum diameter of the tumor was not more than 5cm;
6. Body Mass Index (BMI)≤30kg/m2;
7. No local complications (no obstruction, incomplete obstruction, massive active bleeding, no perforation) Formation of pores and abscesses without invasion of adjacent organs);
8. The hematopoietic functions of heart, lung, liver, kidney and bone marrow meet the requirements of surgery and anesthesia;
9. Voluntarily sign the informed consent form.

Exclusion criteria:

1. Preoperative evaluation of lateral lymph node metastasis;
2. Previous history of malignant tumor;
3. Simultaneous multiple primary colorectal cancer;
4. Patients with contraindications of laparoscopic surgery, such as severe cardiopulmonary insufficiency;
5. Previous multiple abdominal and pelvic surgeries or extensive abdominal adhesions;
6. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc., requiring emergency surgery;
7. Patients with familial adenomatous polyposis, Lynch syndrome associated rectal cancer, and active inflammatory bowel disease;
8. have a history of serious mental illness;
9. pregnant or lactating women;
10. Patients with uncontrolled infection before operation;
11. The investigator did not consider the patient to be eligible for the trial.

Exit Criteria:

1. Patients with distant metastasis confirmed by intraoperative exploration or postoperative pathology, including liver, pelvic cavity, ovary, peritoneum, distant lymph node metastasis, etc.;
2. Intraoperative exploration was necessary for combined organ resection;
3. After enrollment in the study, patients requiring emergency surgical resection due to intestinal obstruction, intestinal perforation, intestinal bleeding, etc.
4. Patients who requested to withdraw from the study cohort for various reasons after enrollment;
5. Those who fail to complete the institute planning for various reasons after being enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were aged between 18 and 75 years;
2. Pathologically confirmed as adenocarcinoma;
3. Colonoscopy or imaging examination confirmed that the distance between the lower edge of the tumor and the anal margin was ≤ 5cm;
4. Preoperative imaging diagnosis was ct1-3nxm0;
5. Preoperative colonoscopy or imaging diagnosis confirmed that the maximum diameter of the tumor was not more than 5cm;
6. Body mass index (BMI) ≤ 30kg / m2;
7. No local complications (no obstruction, incomplete obstruction, no massive active bleeding, no puncture Formation of pores and abscesses without invasion of adjacent organs);
8. The hematopoietic functions of heart, lung, liver, kidney and bone marrow meet the requirements of surgery and anesthesia;
9. Voluntary informed consent.

Exclusion Criteria:

1. Preoperative evaluation of patients with lateral lymph node metastasis;
2. Previous history of malignant tumor;
3. Simultaneous multiple primary colorectal cancer was diagnosed;
4. There are contraindications to laparoscopic surgery, such as severe cardiopulmonary insufficiency;
5. Patients who had undergone abdominal and pelvic surgery for many times or had extensive abdominal adhesions;
6. Patients with intestinal obstruction, intestinal perforation, intestinal hemorrhage and other emergency operations;
7. Patients with familial adenomatous polyposis, Lynch syndrome associated rectal cancer, and inflammatory bowel disease in the active phase;
8. Have a history of serious mental illness;
9. Pregnant or lactating women;
10. Patients with uncontrolled infection before operation;
11. The investigator considered that the patient should not participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival rate | 2-year
  After the postoperative review, the patient had no tumor recurrence and metastasis